CLINICAL TRIAL: NCT02564848
Title: IIT2015-06-Chung: Safety and Efficacy of Omission of Sentinel Node Biopsy in Patients With Clinical T1-2 Estrogen-Positive Breast Cancer Over Age 65
Brief Title: Safety and Efficacy of Omission of Sentinel Node Biopsy in Patients With Estrogen-Positive Breast Cancer Over Age 65
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Alice Chung, Assistant Professor of Surgery, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2015-06-Chung-SNBO
Record Dates: First submitted 2015-09-25; First posted 2015-10-01 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Clinical T1-2N0 ER+; Invasive breast cancer; estrogen-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Segmental; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumpectomy without sentinel node biopsy (Experimental): Subjects will undergo standard of care lumpectomy. A biopsy of the sentinel node will not be performed. After surgery, subjects will receive standard of care radiation on the affected breast and hormonal therapy.
  Interventions: Procedure: Lumpectomy without sentinel node biopsy

INTERVENTIONS:
Procedure: Lumpectomy without sentinel node biopsy — Biopsy of the sentinel node is considered standard of care treatment for women with localized breast cancer. The procedure will be eliminated at time of lumpectomy.

SUMMARY:
This study will examine the outcomes of lumpectomy, surgery to remove a tumor, without sentinel node biopsy (SNB) for women at least 65 years of age with clinically node-negative breast cancer. Clinically node-negative means that during a physical exam your doctor cannot feel or see that any lymph nodes near the breast area are swollen and there is also no imaging evidence, such as from a mammogram, of nodal involvement.

DETAILED DESCRIPTION:
The primary objective of the study is to determine whether omission of sentinel node biopsy in patients who meet eligibility criteria results in an acceptable regional recurrence rate over a 6-year period. A regional recurrence is defined as any recurrence in the ipsilateral axillary nodes, supraclavicular nodes or internal mammary nodes.

Eligible patients will undergo standard of care lumpectomy without sentinel node biopsy followed by radiation and hormonal therapy or have already undergone the procedure prior to enrollment in the study. She may also receive chemotherapy as determined by her treating physician. A physical examination of the affected breast and regional lymph nodes will be conducted every six months for the first two years of follow up and then yearly for the last 3 years of follow up. Imaging of the affected breast will occur every 12 months after surgery per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Female age 65 and older
* Staging:

  1. Patients enrolled prior to surgery: Diagnosis of clinical T1-2N0, ER+, HER2-negative, invasive breast cancer as determined by treating physician. DCIS or LCIS may be present with invasive cancer.
  2. Patients enrolled after surgery: pT1-2NX, or pT1-2N0, ER+, HER2-negative, invasive breast cancer. DCIS or LCIS may be present with invasive cancer.
* Plan to undergo lumpectomy within 3 months of study registration, or underwent lumpectomy within 60 days of study registration (without sentinel node biopsy)
* Patients in whom lymph nodes are palpable and not suspicious who are found to be nodal tumor-free by nodal core needle biopsy are permitted, but those with biopsy-proven nodal metastases are excluded

Exclusion Criteria:

* Patients with diagnosis of ductal or lobular carcinoma in situ
* Patients with diagnosis of inflammatory breast cancer
* Patients who have undergone neoadjuvant chemotherapy for current primary breast cancer (past treatments for other cancers are acceptable)
* Patients planning to have mastectomy or had a mastectomy of the ipsilateral breast
* Prior history of ipsilateral (invasive or DCIS) breast cancer
* Diagnosis of clinical T3 or T4 breast cancer

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-01-22 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Regional recurrence | A regional recurrence during six years of follow-up after lumpectomy.
  A regional recurrence is defined as any recurrence in the ipsilateral axillary nodes, supraclavicular nodes or internal mammary nodes and will be determined by physical exam and breast imaging

SECONDARY OUTCOMES:
Disease-free survival | From date of diagnosis until the date of locoregional or distant recurrence assessed up to 5 years.
Overall survival | From date of diagnosis until the date of death from any cause assessed up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Chung, MD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Chung AP, Dang CM, Karlan SR, Amersi FF, Phillips EM, Boyle MK, Cui Y, Giuliano AE. A Prospective Study of Sentinel Node Biopsy Omission in Women Age >/= 65 Years with ER+ Breast Cancer. Ann Surg Oncol. 2024 May;31(5):3160-3167. doi: 10.1245/s10434-024-15000-w. Epub 2024 Feb 12. PMID 38345718